CLINICAL TRIAL: NCT01248455
Title: A Phase II Trial of IPH2101 (Anti-KIR) in Smoldering Multiple Myeloma (SMM)
Brief Title: A Phase II Trial of Anti-KIR in Smoldering Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients meeting the defined primary obj. (50% decline in M-protein).
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dickran Kazandjian, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110024; 11-C-0024
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma; Myeloma; Smoldering Multiple Myeloma
Keywords: Monoclonal Antibody; NK Cell Mediated Killing; Response Rate; Pharmacokinetics; Biological Activity; Smoldering Multiple Myeloma; SMM
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- anti-KIR in Smoldering Multiple Myeloma Patients (Experimental): Patients will receive anti-KIR(IPH2101) (1mg/kg) every other month for 6 cycles
  Interventions: Drug: (Anti-KIR)

INTERVENTIONS:
Drug: (Anti-KIR) — Patients will receive anti-KIR(IPH2101) (1mg/kg) every other month for 6 cycles

SUMMARY:
Background:

* Recent studies have shown that smoldering multiple myeloma has a high risk of progressing to multiple myeloma, an aggressive type of bone marrow cancer, within 5 years of diagnosis. People with smoldering multiple myeloma have abnormal blood test results that show a high level of monoclonal protein (M-protein) in the blood and of plasma cells in the bone marrow. There are currently no known effective treatments to prevent smoldering multiple myeloma from developing into multiple myeloma, and there are no known tests for determining whether an individual with smoldering multiple myeloma will develop multiple myeloma.
* Certain cells in the immune system, known as natural killer (NK) cells, are active against multiple myeloma. The experimental drug anti-killer cell immunoglobulin-like receptor (anti-KIR) has been shown to help NK cells kill multiple myeloma cells. Researchers are interested in determining whether anti-KIR can be given to individuals with smoldering multiple myeloma to improve their abnormal blood test results.

Objectives:

- To evaluate the safety and effectiveness of anti-KIR as a treatment for abnormal blood test results related to smoldering multiple myeloma.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with smoldering multiple myeloma.

Design:

* Participants will be screened with a physical examination and medical history, and will provide baseline blood, urine, and bone marrow samples before beginning the study drug.
* Participants will receive anti-KIR intravenously for 1 hour, and will be closely monitored for 24 hours after receiving the first dose. If there are no serious side effects, participants will receive five additional anti-KIR doses, one every other month, for a total of six treatment cycles.
* Participants will have monthly visits to provide additional blood and urine samples, and may have additional bone marrow biopsies as directed by the study researchers.
* Participants will have followup visits every 3 to 6 months for up to 5 years after receiving anti-KIR treatment.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is an incurable plasma cell neoplasm with a median survival of 3-4 years.
* Smoldering multiple myeloma (SMM) is a premalignant plasma cell disorder characterized by monoclonal protein greater than or equal to 3 g/dL or bone marrow plasma cells greater than or equal to 10 percent in the absence of myeloma-related tissue impairment with 51 percent progression to MM at 5 years.
* Current recommendations do not endorse treatment of SMM with chemotherapy.
* Transplanted Natural Killer (NK) Cells have anti-myeloma activity.
* Anti-KIR (IPH2101) is a monoclonal antibody that facilitates NK cell mediated killing of myeloma cells by blocking inhibitory receptors (KIR) on NK cells.

Objectives:

* To assess the response rate of anti-KIR(IPH2101) in patients with SMM
* To evaluate the toxicity of anti-KIR(IPH2101) in patients with SMM
* To evaluate the pharmacokinetic parameters and biological activity of anti-KIR (IPH2101)

Eligibility:

* A confirmed diagnosis of SMM
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status in the range of 0-1.
* Without serious co-morbidity that would interfere with receipt of anti-KIR(IPH2101)

Design:

* Single-arm Phase II trial of anti-KIR(IPH2101) for patients with SMM.
* All patients will have initial evaluation and confirmation of diagnosis.
* Patients will receive anti-KIR(IPH2101) (1mg/kg) every other month for 6 cycles.
* Patients will have routine blood work with serum protein electrophoresis (SPEP) and immunofixation monthly.
* Pre- and post-treatment bone marrow biopsies will be obtained for confirmation of diagnosis and correlative studies.
* Patients may donate cellular products or tissues as appropriate for research purposes.
* Optimal two-stage phase II design will be employed, initially enrolling 9 patients. If 3 or more have a positive outcome, then a total of 21 patients will be enrolled in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of smoldering multiple myeloma (SMM) will be made in accordance with the clinical diagnostic criteria set forth by the International Myeloma Working Group. These criteria include:

  * Serum M-protein greater than or equal to 3 g/dl and/or bone marrow plasma cells greater than or equal to 10 percent
  * Absence of anemia: Hemoglobin greater than or equal to 10 g/dl
  * Absence of renal failure: calculated creatinine clearance (according to modification of diet in renal disease (MDRD)) greater than or equal to 40 ml/min (or alternatively based on standard creatinine level criteria of 2 mg/dl)
* Absence of hypercalcemia: Calcium less than or equal to 10.5 mg/dl
* Absence of lytic bone lesion (skeletal survey)
* The diagnoses will be confirmed by serum/urine protein electrophoresis, immunofixation and light-chain assays; as well as immunohistochemical analyses of the bone marrow biopsy.
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Male or female patient who accepts and is able to use recognized effective contraception (oral contraceptives, intrauterine contraceptive device (IUCD), barrier method of contraception in conjunction with spermicidal jelly) through the study and for four months following the final dose of study drug when relevant.
* The patient must be competent to sign an informed consent form.

EXCLUSION CRITERIA:

* Patients with a diagnosis of multiple myeloma (MM) or a clinical suspicion of an ongoing progression into full-blown MM
* Patients without measurable disease defined as serum monoclonal protein (M-protein) less than 1 g/dL.
* Previous treatment having a proven or potential impact on myeloma cell proliferation or survival (including conventional chemotherapies, immunomodulatory drugs (IMiDs), or proteasome inhibitors).
* Use of any investigational agent within the last 3 months.
* Clinical laboratory values at screening:

  * Platelet levels less than 75 times 10^9/L
  * Absolute neutrophil count (ANC) levels less than 1 times 10^9/L
  * Bilirubin levels greater than 1.5 upper limit of normal (ULN) ; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 3.0 ULN (grade 1 National Cancer Institute (NCI))
* Primary or associated amyloidosis
* Known abnormal cardiac status with any of the following:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction within the previous 6 months
  * Symptomatic and/or treatment-refractory cardiac arrhythmia. Patients with controlled or asymptomatic arrhythmia are not excluded from this study.
* Current active infectious disease or positive serology for:

  * Human Immunodeficiency Virus (HIV)
  * Hepatitis C Virus (HCV)
  * Hepatitis B Surface Antigen
* Severe type of autoimmune disease defined as:

  * One which currently requires or previously required long-term systemic immunosuppressive or immunomodulatory therapy (including corticosteroids, administered by systemic route)
  * And/or it has a substantial probability to cause an irreversible injury to any tissue (e.g. Hashimoto thyroiditis).
  * And/or it is recent or unstable, or has a substantial risk to progress and cause severe complications (e.g. Graves disease)
  * Enrollment of other non severe types of auto-immunes disease requiring topical therapy, or non-steroidal inflammatory drugs (NSAIDS) can be considered on a case by case basis by the Principal Investigator.
* History of a lymphoproliferative malignancy.
* History of other malignancy (apart from basal cell carcinoma of the skin or in situ cervical carcinoma) except if the patient has been free of symptoms and without active therapy during at least the previous 5 years.
* Serious concurrent uncontrolled medical disorder.
* History of allograft or solid organ transplantation.
* Any psychological or familial condition potentially interfering with compliance with the study protocol and follow-up schedule.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson KC, Kyle RA, Rajkumar SV, Stewart AK, Weber D, Richardson P; ASH/FDA Panel on Clinical Endpoints in Multiple Myeloma. Clinically relevant end points and new drug approvals for myeloma. Leukemia. 2008 Feb;22(2):231-9. doi: 10.1038/sj.leu.2405016. Epub 2007 Nov 1. PMID 17972944
- [Background] Kristinsson SY, Landgren O, Dickman PW, Derolf AR, Bjorkholm M. Patterns of survival in multiple myeloma: a population-based study of patients diagnosed in Sweden from 1973 to 2003. J Clin Oncol. 2007 May 20;25(15):1993-9. doi: 10.1200/JCO.2006.09.0100. Epub 2007 Apr 9. PMID 17420512
- [Background] Landgren O, Kyle RA, Pfeiffer RM, Katzmann JA, Caporaso NE, Hayes RB, Dispenzieri A, Kumar S, Clark RJ, Baris D, Hoover R, Rajkumar SV. Monoclonal gammopathy of undetermined significance (MGUS) consistently precedes multiple myeloma: a prospective study. Blood. 2009 May 28;113(22):5412-7. doi: 10.1182/blood-2008-12-194241. Epub 2009 Jan 29. PMID 19179464
- [Result] Korde N, Carlsten M, Lee MJ, Minter A, Tan E, Kwok M, Manasanch E, Bhutani M, Tageja N, Roschewski M, Zingone A, Costello R, Mulquin M, Zuchlinski D, Maric I, Calvo KR, Braylan R, Tembhare P, Yuan C, Stetler-Stevenson M, Trepel J, Childs R, Landgren O. A phase II trial of pan-KIR2D blockade with IPH2101 in smoldering multiple myeloma. Haematologica. 2014 Jun;99(6):e81-3. doi: 10.3324/haematol.2013.103085. Epub 2014 Mar 21. No abstract available. PMID 24658821
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0024.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-KIR in Smoldering Multiple Myeloma Patients
Started | 9
Completed | 8
Not Completed | 1
Not completed — switched to alternate treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anti-KIR in Smoldering Multiple Myeloma Patients
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.41 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate is defined as the percentage of participants with a 50% decline in monoclonal protein (M-protein) assessed by the International Multiple Myeloma Working Group (IMWG) for multiple myeloma (MM) criteria. Minimal response (MR) is MR >25% and <50% decrease in M-protein. Biochemical progression (BP) is asymptomatic, ≥ 25% M-protein increase from baseline and an absolute increase of M-protein of 0.75 g/dL demonstrated on two separate occasions. Progressive disease (PD), (clinical progression to symptomatic MM) is development of CRAB (hyperCalcemia (corrected calcium >2.75 mmol/L), Renal insufficiency (attributed to MM), Anemia (hemoglobin <10g/dL), and Bone lesions (lytic lesions or osteoporosis with compression fractures) criteria end organ damage. Stable disease (SD) is not meeting the criteria for minimal response, biochemical progression and progressive disease.
Time Frame: 1 year
Population: Study stopped after the first stage due to the lack of patients meeting the defined primary objective (50% decline in M-protein).
Measure: Number; unit: percentage of participants
Arm/Group | Anti-KIR in Smoldering Multiple Myeloma Patients
Number analyzed (Participants) | 9
percentage of participants
  Minimal Response (MR) | 11
  Stable Disease (SD) | 66
  Biochemical Progression (BP) | 11
  Progressive Disease (PD) | 11
Statistical Analysis 1: Comparison: Anti-KIR in Smoldering Multiple Myeloma Patients; No patients obtained a 50% reduction in M-protein concentration and the study did not continue to the second stage of enrollment due to the lack of efficacy as defined by out criteria. This statistical analysis includes all participants (i.e., stable disease (SD), minimal response (MR), biochemical progression (BP), and progressive disease (PD)); Test type: Superiority or Other; p = 0.56, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Count of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 3 years and 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-KIR in Smoldering Multiple Myeloma Patients
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 3 years and 5 months.
Arm/Group | Anti-KIR in Smoldering Multiple Myeloma Patients
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-KIR in Smoldering Multiple Myeloma Patients (N=9)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (11)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CPK increased (Investigations) | 2 (6)
Chills (General disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Flashing lights (Eye disorders) | 1 (2)
Floaters (Eye disorders) | 1 (1)
Flu like symptoms (General disorders) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (8)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (22)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (9)
Hypothyroidism (Endocrine disorders) | 1 (2)
Lymphocyte count decreased (Investigations) | 6 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other, carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Platelet count decreased (Investigations) | 3 (8)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, scalp lesion/scab (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 5 (16)

LIMITATIONS AND CAVEATS:
Study stopped after the first stage due to lack of patients meeting the defined primary objective (50% decline in M-protein). The study did not continue to the second stage of enrollment due to lack of efficacy as defined by our criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2013-03-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT01248455/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT01248455/Prot_SAP_002.pdf